CLINICAL TRIAL: NCT04178629
Title: Characterization of Ceftobiprole's Cerebrospinal Fluid Penetration in Patients With External Ventricular Derivation
Brief Title: Ceftobiprole's Cerebrospinal Fluid Penetration in Patients With External Ventricular Derivation (CEFTO-EVD)
Acronym: CEFTO-EVD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Collaborators: University of Turin, Italy (Other); University of Pisa (Other); Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Piva Simone, Assistant Professor, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Other Study IDs: NP3617
Record Dates: First submitted 2019-10-15; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Pharmacokinetics; Cerebral Ventriculitis; Cephalosporins; Cerebrospinal Fluid
Keywords: Ceftobiprole; External Ventricular Derivation; Cerebrospinal fluid penetration; ATP Binding Cassette Transporter, Subfamily B, Member 1; Tissue Distribution
MeSH Terms: conditions — Cerebral Ventriculitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Serum
  * Cerebrospinal Fluid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Cerebrospinal fluid penetration of ceftobiprole has been studied in an animal model of meningitidis. Ceftobiprole is bactericidal, well tolerated and it has anti-biofilm activity. Altogether, these pharmacodynamics and pharmacokinetic properties of ceftobiprole are suitable for its use in case of External Ventricular Derivation(EVD)-related ventriculitis. Nowadays there are no human studies on the penetration and efficacy of ceftobiprole in the CSF. The study aims to evaluate characteristics of the CSF penetration of Ceftobiprole after intravenous administration in patients with EVD, that need for a concomitant infection this therapy (prescribed by an Infectious Diseases doctor).

DETAILED DESCRIPTION:
According with Inclusion and Exclusion criteria, patients with an EVD and concomitant ceftobiprole therapy will be enrolled in the study.

In particular, ceftobiprole will be prescribed by an expert infectivologist, in accordance with the MHRA guidelines.

Once the patients will be enrolled, Ceftobiprole will be administered by 2 hr i.v. infusion at the following dosage:

* normal renal function: 500mg every 8 hr
* mild renal impairment (50-80mL/min): 500mg every 8 hours
* moderate (30-49mL/min): 500mg every 12 hours
* severe (<30mL/min): 250mg every 12 hours.

The following blood and CSF sample will be drowned only during the third dose of antibiotic therapy. Blood Samples (1 mL each) will be obtained at the following time points: before and at the end of infusion of ceftobiprole, then 0.5, 1, 2, 2.5, 3 and 4 hr after drug administration (total of 8 samples), using a single venous or arterial line cannulation. CSF samples: 0.5ml will be drawned from implanted EVD with a sterile field at the same blood sample time-point, and at 6, 8 and 10 hr after the end of drug administration (11 samples total).

CSF and blood will be spin-down at 3000 rpm for 10 minutes and then stored at -80°C.

Samples will be sent all in once by courier to Laboratory of Clinical Pharmacology and Pharmacogenetics, University of Turin, Department of Medical Sciences, Amedeo di Savoia Hospital, Turin (Italy) in order to determine the serum and CSF concentration.

Ceftobiprole concentrations (both in plasma/serum and CFS) will be analyzed with EMA validated LC-MS/MS methods.

MDR1 gene polymorphisms will be analyzed with RT-PCR instrument, using commercial genetic probes on the blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Age>18
* Patients with External Ventricular Derivation (EVD)
* Patients who receive ceftobiprole for any infection where Ceftobiprole could be used, as judged by an expert infectivologist
* Patients or their relatives/parents who consent to study participation

Exclusion Criteria:

* Patients with end-stage renal insufficiency
* Patients with a BMI>30
* Pregnancy
* Moribund patients
* Allergy to cephalosporine or ceftobiprole
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient admitted in Intensive Care Unit or Neurosurgical Unit of Hospital "Spedali Civili di Brescia" (BS, Italy), according to Inclusion and Exclusion Criteria, with an EVD and concomitant Ceftobiprole therapy. When ceftobiprole will be administered i.v. for the first time, patients will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2019-07-02 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Ceftobiprole's CSF penetration | Blood samples: before infusion, end of infusion, then 30 minutes, 1 hour, 2 hours, 2,5 hours, 3 hours, 4 hours after end of administration; CSF samples: at the same time of blood samples, then at 6 hours, 8 hours and 10 hours after end of administration
  Evaluate the Cerebrospinal Fluid penetration of Ceftobiprole in patients with External Ventricular Derivation. Ceftobiprole concentrations (both in plasma/serum and CFS) will be analyzed with EMA fully validated LC-MS/MS methods.

SECONDARY OUTCOMES:
Ceftobiprole's MDR1 role | The MDR1 gene will be analyzed on whole blood samples, by real-time PCR, through study completion, an average of 18 months.
  Evaluate the role of MDR1 polymorphisms in modulating ceftobiprole CSF penetration.
Ceftobiprole's efficacy in CSF | The measurement is assessed through study completion, an average of 18 months.
  In vitro, the efficacy of ceftobiprole against the most common pathogen causing Ventricular Meningitis (MRSA, MRSE, Pseudomonas Aeruginosa and Enterobacteriaceae) will be assessed using the percentage of time during which the free CSF ceftobiprole concentration remains above the minimal inhibitory concentration (MIC)

CONTACTS AND LOCATIONS:
Overall Officials: Simone Piva, Principal Investigator — Università degli Studi di Brescia
Locations (1):
- Spedali Civili di Brescia, Brescia, Italy

IPD SHARING:
Plan to Share IPD: Yes
The database is in RedCap. We could share all data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: already available